CLINICAL TRIAL: NCT02054689
Title: PHASE I STUDY OF FRACTIONATED STEREOTACTIC RADIOSURGERY FOR LARGE BRAIN METASTASES
Brief Title: Fractionated Stereotactic Radiosurgery for Large Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven Burton (Other)
Responsible Party: Sponsor-Investigator, Steven Burton, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 11-091
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Large Brain Mets
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fractionated Stereotactic Radiosurgery (Other): 24 to 36 Gy in 3 fractions (8-12 Gy/fx).
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Fractionated Stereotactic Radiosurgery — SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
  Other Names: SRS; SBRT; CyberKnife; Trilogy; True Beam; Radiosurgery

SUMMARY:
This is a research trial that seeks to break up the total radiation dose into multiple smaller radiation treatments, termed fractionated stereotactic radiosurgery (FSRS) which may make the treatment feasible. Fractionated sterotatcic radiation, the risks of FSRS, and possible costs will be described later in this document. This clinical trial is for people who have had no prior whole brain radiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* A life expectancy of at least 12 weeks with a Karnofsky performance status of at least 70 (Appendix II)
* The target lesion(s) can be accurately measured in at least one dimension according to RECIST
* No prior radiotherapy to the brain
* Previous or concurrent systemic or targeted chemotherapy is allowed
* Patients must have an extra-cranial primary tumor diagnosis
* Patients will have no more than 3 distinct lesions within the brain. At least 1 lesion must be a minimum of 3cm in greatest dimension, no larger than 5cm which will be treatable by fractionated stereotactic radiosurgery
* The additional lesions will each be treated with single fraction stereotactic radiosurgery
* Patient may be on steroids or anti-epileptics
* Must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts
* Patients do not need a histologically proven diagnosis of brain mets

Exclusion Criteria:

* Symptomatic patients in need of surgery to the "target" lesion
* Four or more newly-diagnosed lesions
* Prior surgical resection of targeted tumor
* Prior WBRT
* Primary brain tumor
* Pregnant or breast-feeding patients
* Primary tumor histology of lymphoma, leukemia, multiple myeloma or germ cell tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burton, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fractionated Stereotactic Radiosurgery - 24Gy: 24 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 27Gy: 27 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 30 Gy: 30 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 33 Gy: 33 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 36 Gy: 36 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam
Period: Overall Study
Arm/Group | Fractionated Stereotactic Radiosurgery - 24Gy | Fractionated Stereotactic Radiosurgery - 27Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Started | 4 | 2 | 3 | 2 | 9
Completed | 4 | 2 | 3 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fractionated Stereotactic Radiosurgery - 24 Gy: 24 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 27 Gy: 27 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Fractionated Stereotactic Radiosurgery - 36 Gy: 36 Gy in 3 fractions (8-12 Gy/fx).
  Fractionated Stereotactic Radiosurgery: SRS SBRT CyberKnife Trilogy True Beam Radiosurgery
- Total: Total of all reporting groups
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy | Total
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9 | 20
Age, Continuous [Median (Full Range); unit: years] | 69.5 [53.0 to 89.0] | 66.5 [56.0 to 77.0] | 54.0 [46.0 to 70.0] | 61.5 [40.0 to 83.0] | 65.0 [43.0 to 87.0] | 67.0 [40.0 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 7 | 14
  Male | 2 | 1 | 0 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 3 | 2 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 4 | 2 | 3 | 1 | 7 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing DLT
Description: The number of patients experiencing DLT, defined as the maximum amount of Gy fractionated stereotactic radiosurgery (FSRS) delivered without significant toxicity.
Time Frame: Up to 3 years
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9
participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was determined following a Time-to-Event Continual Reassessment Model which models toxicity as a function of dose. Treatment was given in 3 fractions (8-12 Gy/fx).
Time Frame: Up to 24 months post completion of treatment
Population: All treated patients evaluable for DLTs
Measure: Number; unit: Gy
Groups:
- All Participants: An evaluable patient is defined as one who either a) completes the three fractions and has no DLT until one month after the last fraction, or b) a patient who received at least one fraction and suffers DLT.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Gy | 36

3. Secondary Outcome: Best Response
Description: Percentage of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) in the target lesion, or Progressive Disease (PD) per RECIST v1.1. (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. (PR): at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. (PD): at least a 20% increase in the sum of diameters of target lesions, taking as a reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 24 months after completion of treatment
Population: Treated patients who were radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 1 | 0 | 2
  Stable Disease | 1 | 0 | 1 | 0 | 3
  Progressive Disease | 3 | 1 | 1 | 2 | 4

4. Secondary Outcome: Local Control of Disease
Description: Percentage of patients with local control, defined as stable disease (SD), partial response (PR), or complete response (CR) in the target lesion, per RECIST v1.1. Complete Response (CR): the disappearance of a target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm., Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 24 months after completion of treatment
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9
percentage of participants
  Local Control - Yes | 25 | 50 | 66.7 | 0 | 55.6
  Local Control - No | 75 | 50 | 33.3 | 100 | 44.4

5. Secondary Outcome: Regional Intracranial Failure
Description: Percentage of patients who develop new lesions outside the target volume. Patients without follow-up scans are excluded as it is not known if they developed lesions outside the target volume.
Time Frame: Up to 24 months after completion of treatment
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9
percentage of patients
  Yes | 25 | 100 | 66.7 | 0 | 22.2
  Unknown - no FU scans | 25 | 0 | 0 | 50 | 22.2
  No | 50 | 0 | 33.3 | 50 | 55.6

6. Secondary Outcome: Functional Assessment of Cancer Therapy - Brain (FACT-Br)
Description: Functional Assessment of Cancer Therapy - Brain (FACT-Br) is a 50 item, self-administered questionnaire used to assess Quality of Life, including, Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Subscale scores range from 0-4. FACT-G = (PWB - 7 items, score range 0-28) + (SWB - 7 items, score range 0-28) + (EWB - 6 items, score 0-24) + (FWB - 7 items, 0-28). The assessment takes 10-15 minutes to completed and is scored using a 5-point Likert-type scale. Scores range from 0-108, with higher scores indicating better Quality of Life.
Time Frame: Prior to treatment; 30 days post treatment; 8 -12 weeks, 22-28 weeks, 30-42 weeks, 45-60 weeks, 64-74 weeks, 80-84 weeks, 90-96 weeks,100-112 weeks, 120-124 weeks, 130-140 weeks, 145-155 weeks, and 160-170 weeks post treatment
Population: All participants who provided self-administered QoL surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 9
score on a scale
  Prior to treatment: number analyzed (Participants) | 4 | 2 | 2 | 2 | 7
  Prior to treatment | 76 (21) | 83 (13) | 76 (12) | 59 (25) | 77 (14)
  30 days post treatment: number analyzed (Participants) | 3 | 2 | 1 | 0 | 4
  30 days post treatment | 82 (9) | 79 (18) | 76 (NA) — insufficient number of participants with completed QoL assessment |  | 79 (23)
  8-16 weeks post treatment: number analyzed (Participants) | 3 | 2 | 2 | 0 | 2
  8-16 weeks post treatment | 81 (14) | 84 (5) | 83 (2) |  | 87 (10)
  22-28 weeks post treatment: number analyzed (Participants) | 2 | 0 | 2 | 0 | 1
  22-28 weeks post treatment | 85 (14) |  | 78 (2) |  | 78 (NA) — insufficient number of participants with completed QoL assessment
  30-42 weeks post treatment: number analyzed (Participants) | 2 | 1 | 2 | 0 | 1
  30-42 weeks post treatment | 90 (11) | 92 (NA) — insufficient number of participants with completed QoL assessment | 85 (6) |  | 59 (NA) — insufficient number of participants with completed QoL assessment
  45-60 weeks post treatment: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0
  45-60 weeks post treatment | 98 (NA) — insufficient number of participants with completed QoL assessment | 94 (NA) — insufficient number of participants with completed QoL assessment | 83 (NA) — insufficient number of participants with completed QoL assessment |  |
  64-74 weeks post treatment: number analyzed (Participants) | 1 | 1 | 1 | 0 | 1
  64-74 weeks post treatment | 95 (NA) — insufficient number of participants with completed QoL assessment | 101 (NA) — insufficient number of participants with completed QoL assessment | 62 (NA) — insufficient number of participants with completed QoL assessment |  | 79 (NA) — insufficient number of participants with completed QoL assessment
  80-84 weeks post treatment: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0
  80-84 weeks post treatment |  | 102 (NA) — insufficient number of participants with completed QoL assessment | 64 (NA) — insufficient number of participants with completed QoL assessment |  |
  90-96 weeks post treatment: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  90-96 weeks post treatment |  | 90 (NA) — insufficient number of participants with completed QoL assessment |  |  |
  100-112 weeks post treatment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  100-112 weeks post treatment | 98 (NA) — insufficient number of participants with completed QoL assessment |  |  |  |
  120-124 weeks post treatment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  120-124 weeks post treatment | 104 (NA) — insufficient number of participants with completed QoL assessment |  |  |  |
  130-140 weeks post treatment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  130-140 weeks post treatment | 106 (NA) — insufficient number of participants with completed QoL assessment |  |  |  |
  145-155 weeks post treatment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  145-155 weeks post treatment | 100 (NA) — insufficient number of participants with completed QoL assessment |  |  |  |
  160-170 weeks post treatment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  160-170 weeks post treatment | 99 (NA) — insufficient number of participants with completed QoL assessment |  |  |  |

ADVERSE EVENTS:
Time Frame: Adverse Events data collected for a total of 10 years for the study population. Up to approximately 24 months after start of treatment for individuals.
Arm/Group | Fractionated Stereotactic Radiosurgery - 24 Gy | Fractionated Stereotactic Radiosurgery - 27 Gy | Fractionated Stereotactic Radiosurgery - 30 Gy | Fractionated Stereotactic Radiosurgery - 33 Gy | Fractionated Stereotactic Radiosurgery - 36 Gy
All-Cause Mortality (participants affected / at risk) | 4/4 | 1/2 | 3/3 | 2/2 | 8/9
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/2 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/4 | 2/2 | 3/3 | 2/2 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fractionated Stereotactic Radiosurgery - 24 Gy (N=4) | Fractionated Stereotactic Radiosurgery - 27 Gy (N=3) | Fractionated Stereotactic Radiosurgery - 30 Gy (N=2) | Fractionated Stereotactic Radiosurgery - 33 Gy (N=3) | Fractionated Stereotactic Radiosurgery - 36 Gy (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fractionated Stereotactic Radiosurgery - 24 Gy (N=4) | Fractionated Stereotactic Radiosurgery - 27 Gy (N=2) | Fractionated Stereotactic Radiosurgery - 30 Gy (N=3) | Fractionated Stereotactic Radiosurgery - 33 Gy (N=2) | Fractionated Stereotactic Radiosurgery - 36 Gy (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0 | 2
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 2 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, specifythrush (General disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, specifylymphadenopathy (General disorders) | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 1 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 1 | 6
Edema limbs (General disorders) | 2 | 0 | 1 | 2 | 4
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, specifyThrush (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 4
Musculoskeletal and connective tissue disorder - Other, specifyrhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specifyBursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, specifyPositive Romberg Sign (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 2
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 1 | 1 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specifyNocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT02054689/Prot_SAP_000.pdf